CLINICAL TRIAL: NCT00500175
Title: Novel Home Care Device for High-Risk Diabetic Patients
Acronym: TempTouchRM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Diabetica Solutions Inc. (Industry)
Collaborators: National Institutes of Health (NIH) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: DK061815
Record Dates: First submitted 2007-07-10; First posted 2007-07-12 (Estimated); Last update posted 2007-07-12 (Estimated); Status verified 2007-07

CONDITIONS: Diabetes; Neuropathic Limb; Elevated Temperature; Shear Pressure; Increased Temperatures
Keywords: diabetes; ulceration; amputation; pressure sores; shear friction
MeSH Terms: conditions — Diabetes Mellitus; Fever; Ulcer; Pressure Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: TempTouchRM
Device: Offloading

SUMMARY:
More than half of all lower extremity amputations are in persons with diabetes. These patients suffer from severe, diabetes-induced, peripheral, sensory neuropathy and, thus they frequently do not protect their feet from repetitive shear stress or traumatic episodes and ulceration often ensues. We have previously shown that the temperature profile of the plantar aspects of the foot provides a reliable warning of tissue injury and can be effectively used as a preventive modality. In this study we propose to further develop and clinically test a novel infrared-based temperature instrument (TempTouchRM®) that is intended for home use by high-risk diabetic patients. This step-on remote monitoring device will serve as an early warning system for impending ulcers and Charcot fractures. The study's central hypothesis is that the TempTouchRM device will reduce the incidence of ulcers by providing an accurate, simple, and effective approach to monitor changes in foot temperatures.

DETAILED DESCRIPTION:
The study's central hypothesis is that the TempTouchRM device will reduce the incidence of ulcers by providing an accurate, simple, and effective approach to monitor changes in foot temperatures. To study this hypothesis, the following specific aims are proposed:

Aim 1: To develop, validate and implement software and protocols for the following: (i) data acquisition and processing, and (ii) the physician-TempTouchRM communications interface. A state-of-the-art web interface will be developed to allow clinicians to view the stored data for their patients.

Aim 2: To evaluate the effectiveness of the TempTouchRM in reducing the incidence of diabetic foot ulcers among high-risk patients. Our hypothesis is that patients monitored with the TempTouchRM will have fewer foot ulcers and that the ulcers will be less severe. The 110 patient study will comprise two treatment arms: the standard therapy group and the enhanced therapy group The latter will receive standard care plus infrared temperature monitoring using the TempTouchRM daily for 12 months. Elevated temperatures will provide information to the physician that prevention practices should be initiated, such as off-loading, skin care, etc.

Aim 3: To determine the normal range of temperature variations for each individual foot for patients in the Enhanced Therapy and to correlate deviations from this range to the incidence of ulcers. Our previous studies have used the contralateral foot as the control to detect abnormal temperatures. We will investigate the hypothesis that with proper trending of normal foot temperatures, the individual foot can serve as its own control for predicting ulcers.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of diabetes by WHO criteria, ability to provide informed consent, 18-80 years of age.

Exclusion Criteria:

* patients with open ulcers or open amputation sites, active Charcot arthropathy, severe peripheral vascular disease, active foot infection, dementia, impaired cognitive function, history of drug or alcohol abuse within one year of the study, or other conditions based on the PI's clinical judgment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2007-01; Study Completion 2008-06 (Estimated)

PRIMARY OUTCOMES:
incident foot ulcers | one year

SECONDARY OUTCOMES:
temperature spikes on foot zones | one year

CONTACTS AND LOCATIONS:
Overall Officials: Kevin R Higgins, DPM, Principal Investigator
Locations (1):
- Kevin R. Higgins, DPM, San Antonio, Texas, United States